CLINICAL TRIAL: NCT04395521
Title: A Facebook Group-based Program for Foot Self-management Support of Adults With Diabetes Mellitus: A Feasibility Study in Canada
Brief Title: The Feasibility of a Facebook Group-based Program for Foot Self-management Support of Adults With Diabetes in Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Obilor (Other)
Collaborators: Wounds Canada (Unknown)
Responsible Party: Sponsor-Investigator, Helen Obilor, Principal investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6029718
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Patient education; Foot self-care; Foot self-care adherence; Social media; Self-management support
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Access to a diabetic foot self-management support program via a Facebook group platform for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook group arm (Experimental): Access to a diabetic foot self-management support program via a Facebook group platform for three months plus the standard care.
  Interventions: Behavioral: Diabetic foot self-management support
- Standard care arm (No Intervention): Carry on with the routine diabetes care offered to the participants in their health facilities.

INTERVENTIONS:
Behavioral: Diabetic foot self-management support — Daily educational organic or inorganic posts (2 to 5) released in a timed sequence through a Hootsuite application plus peer interactions/support for three months.
  Arms: Facebook group arm

SUMMARY:
The primary objective of this study is to examine the feasibility of a Facebook group-based program to support adults with diabetes in their foot self-care and prevention of foot ulcers.

The sub-objectives are:

1. To determine the recruitment and retention rate of participants in the study. 2. To assess the acceptability of the Facebook group program among participants. 3. To determine the level and pattern of engagement by the participants within the Facebook group platform. 4. To determine the efficacy of the Facebook group program and how it works to improve diabetic foot care-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type I or II diabetes;
* 18 years of age or older
* reside in Canada
* Proficiency in the English language - understanding, speaking, reading, and writing.
* Have an active Facebook account or willing to create one
* Have access to the internet and computer or smartphone

Exclusion Criteria:

* Declined consent
* Did not provide follow-up contact information
* Completed less than 60% of the baseline survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
The number of participants that accepted the intervention. | Four weeks after the commencement of intervention.
  Number of participants who scored above 70 in the questionnaire on acceptance and satisfaction with the Facebook group-based program.
The level of participants' engagement in the Facebook group. | Throughout the intervention period (3 months).
  The number of participants who viewed and reacted (comments and likes) to educational posts.
The efficacy of the study intervention on participants' foot self-care adherence. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention foot self-care adherence. Foot self-care adherence will be assessed using an adapted Foot Self-Care Behavior Tool, which consists of 17 items on preventive and potentially destructive foot self-care practices with a score range of 0 - 87.

SECONDARY OUTCOMES:
The efficacy of the study intervention on participants' foot self-care confidence. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention foot self-care confidence. Foot self-care confidence will be measured using the Foot Care Confidence Scale (FCCS), which consists of 12 items on a five-point Likert scale with a score range of 12 - 60.
The efficacy of the study intervention on participants' perceived foot health status. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention perceived foot health status. Perceived foot health status will be assessed using the general foot health questions 9 and 12 of the Foot Health Status Questionnaire with a score range of 2 - 10.
The efficacy of the study intervention on participants' awareness of community resources. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention awareness of community resources. Participants' awareness of community resources will be assessed by asking them to rate the extent to which they can successfully locate available resources in their community for preventing DFU on a scale of 0 - 10.
The efficacy of the study intervention on participants' communication with health care professionals. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention communication with health care professionals. Participants' level of communication with health care professionals about their foot health will be assessed using an adapted Stanford University Chronic Disease Self-Management Program Communication with Physicians' Tool with a score range of 0 - 15.
The efficacy of the study intervention on participants' quality of life. | Two time points > Baseline and at the end of the intervention period (3 months).
  Mean difference in participants' baseline and three-month post-intervention quality of life score. The participants' quality of life will be assessed using the Medical Outcome Study Short Form questionnaire (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Helen N Obilor, MSc., Principal Investigator — Faculty of Health Sciences\School of Nursing, Queen's University; Kevin Woo, Ph.D., Study Director — Faculty of Health Sciences\School of Nursing, Queen's University; Rosemary Wilson, Ph.D., Study Director — Faculty of Health Sciences\School of Nursing, Queen's University; Joan E Tranmer, Ph.D, Study Director — Faculty of Health Sciences\School of Nursing, Queen's University
Locations (1):
- School of Nursing, Queens University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abedin T, Ahmed S, Al Mamun M, Ahmed SW, Newaz S, Rumana N, Turin TC. YouTube as a source of useful information on diabetes foot care. Diabetes Res Clin Pract. 2015 Oct;110(1):e1-e4. doi: 10.1016/j.diabres.2015.08.003. Epub 2015 Aug 13. PMID 26303266
- [Background] Abedin T, Al Mamun M, Lasker MAA, Ahmed SW, Shommu N, Rumana N, Turin TC. Social Media as a Platform for Information About Diabetes Foot Care: A Study of Facebook Groups. Can J Diabetes. 2017 Feb;41(1):97-101. doi: 10.1016/j.jcjd.2016.08.217. PMID 28126155
- [Background] Adarmouch L, Elyacoubi A, Dahmash L, El Ansari N, Sebbani M, Amine M. Short-term effectiveness of a culturally tailored educational intervention on foot self-care among type 2 diabetes patients in Morocco. J Clin Transl Endocrinol. 2017 Feb 9;7:54-59. doi: 10.1016/j.jcte.2017.01.002. eCollection 2017 Mar. PMID 29067251
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Bilandzic A, Rosella L. The cost of diabetes in Canada over 10 years: applying attributable health care costs to a diabetes incidence prediction model. Health Promot Chronic Dis Prev Can. 2017 Feb;37(2):49-53. doi: 10.24095/hpcdp.37.2.03. PMID 28273040
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Bus SA, van Netten JJ. A shift in priority in diabetic foot care and research: 75% of foot ulcers are preventable. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:195-200. doi: 10.1002/dmrr.2738. PMID 26452160
- [Background] Dorresteijn JA, Kriegsman DM, Assendelft WJ, Valk GD. Patient education for preventing diabetic foot ulceration. Cochrane Database Syst Rev. 2014 Dec 16;2014(12):CD001488. doi: 10.1002/14651858.CD001488.pub5. PMID 25514250
- [Background] Fan L, Sidani S, Cooper-Brathwaite A, Metcalfe K. Improving foot self-care knowledge, self-efficacy, and behaviors in patients with type 2 diabetes at low risk for foot ulceration: a pilot study. Clin Nurs Res. 2014 Dec;23(6):627-43. doi: 10.1177/1054773813491282. Epub 2013 Jul 3. PMID 23823459
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Gershater MA, Pilhammar E, Apelqvist J, Alm-Roijer C. Patient education for the prevention of diabetic foot ulcers. European Diabetes Nursing. 2011: 8: 102-107b.
- [Background] Grady PA, Gough LL. Self-management: a comprehensive approach to management of chronic conditions. Am J Public Health. 2014 Aug;104(8):e25-31. doi: 10.2105/AJPH.2014.302041. Epub 2014 Jun 12. PMID 24922170
- [Background] Jeffcoate W, Barron E, Lomas J, Valabhji J, Young B. Using data to tackle the burden of amputation in diabetes. Lancet. 2017 Oct 21;390(10105):e29-e30. doi: 10.1016/S0140-6736(17)32401-7. Epub 2017 Sep 11. No abstract available. PMID 28911921
- [Background] Jeffcoate WJ, Vileikyte L, Boyko EJ, Armstrong DG, Boulton AJM. Current Challenges and Opportunities in the Prevention and Management of Diabetic Foot Ulcers. Diabetes Care. 2018 Apr;41(4):645-652. doi: 10.2337/dc17-1836. PMID 29559450
- [Background] Lincoln NB, Radford KA, Game FL, Jeffcoate WJ. Education for secondary prevention of foot ulcers in people with diabetes: a randomised controlled trial. Diabetologia. 2008 Nov;51(11):1954-61. doi: 10.1007/s00125-008-1110-0. Epub 2008 Aug 30. PMID 18758747
- [Background] Maydick DR, Acee AM. Comorbid Depression and Diabetic Foot Ulcers. Home Healthc Now. 2016 Feb;34(2):62-7. doi: 10.1097/NHH.0000000000000340. PMID 26835804
- [Background] McGowan PT. Self-management education and support in chronic disease management. Prim Care. 2012 Jun;39(2):307-25. doi: 10.1016/j.pop.2012.03.005. Epub 2012 Apr 24. PMID 22608868
- [Background] Monami M, Longo R, Desideri CM, Masotti G, Marchionni N, Mannucci E. The diabetic person beyond a foot ulcer: healing, recurrence, and depressive symptoms. J Am Podiatr Med Assoc. 2008 Mar-Apr;98(2):130-6. doi: 10.7547/0980130. PMID 18347122
- [Background] Monami M, Zannoni S, Gaias M, Nreu B, Marchionni N, Mannucci E. Effects of a Short Educational Program for the Prevention of Foot Ulcers in High-Risk Patients: A Randomized Controlled Trial. Int J Endocrinol. 2015;2015:615680. doi: 10.1155/2015/615680. Epub 2015 Sep 10. PMID 26448748
- [Background] Moorhead SA, Hazlett DE, Harrison L, Carroll JK, Irwin A, Hoving C. A new dimension of health care: systematic review of the uses, benefits, and limitations of social media for health communication. J Med Internet Res. 2013 Apr 23;15(4):e85. doi: 10.2196/jmir.1933. PMID 23615206
- [Background] Obilor HN, Adejumo PO. Assessment of diabetic foot ulcer-related pain and its relationship to quality of life. Wound Practice and Research. 2015; 23 (3): 124-131.
- [Background] Ogrin R, Viswanathan R, Aylen T, Wallace F, Scott J, Kumar D. Co-design of an evidence-based health education diabetes foot app to prevent serious foot complications: a feasibility study. Practical Diabetes. 2018; 35: 203-209d.
- [Background] Partridge SR, Gallagher P, Freeman B, Gallagher R. Facebook Groups for the Management of Chronic Diseases. J Med Internet Res. 2018 Jan 17;20(1):e21. doi: 10.2196/jmir.7558. PMID 29343460
- [Background] Patel R, Chang T, Greysen SR, Chopra V. Social Media Use in Chronic Disease: A Systematic Review and Novel Taxonomy. Am J Med. 2015 Dec;128(12):1335-50. doi: 10.1016/j.amjmed.2015.06.015. Epub 2015 Jul 6. PMID 26159633
- [Background] Petrovski G, Zivkovic M. Impact of Facebook on Glucose Control in Type 1 Diabetes: A Three-Year Cohort Study. JMIR Diabetes. 2017 Jun 7;2(1):e9. doi: 10.2196/diabetes.7693. PMID 30291064
- [Background] Schaper NC, Van Netten JJ, Apelqvist J, Lipsky BA, Bakker K; International Working Group on the Diabetic Foot. Prevention and management of foot problems in diabetes: a Summary Guidance for Daily Practice 2015, based on the IWGDF Guidance Documents. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:7-15. doi: 10.1002/dmrr.2695. PMID 26335366
- [Background] Ahmad Sharoni SK, Abdul Rahman H, Minhat HS, Shariff-Ghazali S, Azman Ong MH. The effects of self-efficacy enhancing program on foot self-care behaviour of older adults with diabetes: A randomised controlled trial in elderly care facility, Peninsular Malaysia. PLoS One. 2018 Mar 13;13(3):e0192417. doi: 10.1371/journal.pone.0192417. eCollection 2018. PMID 29534070
- [Background] Ahmad Sharoni SK, Minhat HS, Mohd Zulkefli NA, Baharom A. Health education programmes to improve foot self-care practices and foot problems among older people with diabetes: a systematic review. Int J Older People Nurs. 2016 Sep;11(3):214-39. doi: 10.1111/opn.12112. Epub 2016 Feb 25. PMID 26916809
- [Background] Smith PE, McGuire J, Falci M, Poudel DR, Kaufman R, Patterson MA, Pelleschi B, Shin E. Analysis of YouTube as a Source of Information for Diabetic Foot Care. J Am Podiatr Med Assoc. 2019 Mar;109(2):122-126. doi: 10.7547/16-149. PMID 31135201
- [Background] Tickle-Degnen L. Nuts and bolts of conducting feasibility studies. Am J Occup Ther. 2013 Mar-Apr;67(2):171-6. doi: 10.5014/ajot.2013.006270. PMID 23433271
- [Background] Torgerson DJ, Sibbald B. Understanding controlled trials. What is a patient preference trial? BMJ. 1998 Jan 31;316(7128):360. doi: 10.1136/bmj.316.7128.360. No abstract available. PMID 9487173
- [Background] Ventola CL. Social media and health care professionals: benefits, risks, and best practices. P T. 2014 Jul;39(7):491-520. PMID 25083128
- [Background] Woo K. New initiative: Online social support program for people with diabetes and foot ulcers. Diabetic Foot Canada. 2014; 2(3): 11-12.
- [Background] Woodbury MG, Botros M, Kuhnke JL, Greene J. Evaluation of a peer-led self-management education programme PEP Talk: Diabetes, Healthy Feet and You. Int Wound J. 2013 Dec;10(6):703-11. doi: 10.1111/iwj.12188. PMID 26074389
- [Derived] Obilor HN, Veryha O, Weisz T, Botros M, Wilson R, Tranmer J, Woo K. The feasibility of a social media-based foot self-management education and support program for adults with diabetes: A partially randomized preference trial. PEC Innov. 2024 Jun 18;5:100307. doi: 10.1016/j.pecinn.2024.100307. eCollection 2024 Dec 15. PMID 39027228
- See also: Foundations of best practice for skin and wound management: Best practice recommendations for the prevention and management of diabetic foot ulcers — http://www.woundscanada.ca/docman/public/health-care-professional/bpr-workshop/895-wc-bpr-prevention-and-management-of-diabetic-foot-ulcers-1573r1e-final/file
- See also: The economic impact of offloading devices for the prevention of amputations in Ontario. — http://www.diabetes.ca/advocacy---policies/advocacy-reports/amputation-prevention-reports
- See also: Share of U.S. adults using social media, including Facebook, is mostly unchanged since 2018 — http://www.pewresearch.org/fact-tank/2019/04/10/share-of-u-s-adults-using-social-media-including-facebook-is-mostly-unchanged-since-2018/
- See also: Clinical best practice guidelines: Assessment and management of foot ulcers for people with diabetes. — http://rnao.ca/sites/rnao-ca/files/Assessment_and_Management_of_Foot_Ulcers_for_People_with_Diabetes_Second_Edition1.pdf
- See also: IWGDF Practical Guidelines on the Prevention and Management of Diabetic Foot Disease. — http://iwgdfguidelines.org/wp-content/uploads/2019/05/01-IWGDF-practical-guidelines-2019.pdf
- See also: Most popular social networks worldwide as of October 2019, ranked by number of active users. — http://www.statista.com/statistics/272014/global-social-networks-ranked-by-number-of-users/
- See also: Social Networking in Canada. — http://www.statista.com/study/32357/social-networking-in-canada-statista-dossier/
- See also: Diabetes-prevalence and care practices: Findings. — https://www150.statcan.gc.ca/n1/pub/82-003-x/2008003/article/10663/5202464-eng.htm